CLINICAL TRIAL: NCT06552286
Title: A Multisite RCT of a Daily Living Skills Intervention for Autistic Adolescents Prior to the Transition to Adulthood
Brief Title: STRW-T Intervention for Autistic Adolescents in 11th and 12th Grade
Acronym: STRW-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN-DUNCAN-2023-0476; 1R01HD113529-01 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial - A study in which the participants are divided by chance into separate groups that compare different treatments or other interventions.
Who Masked: Outcomes Assessor
Masking Description: Coordinator who is assessing goals of participants is masked from knowing which group each participant was randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surviving and Thriving in the Real World - Telehealth (STRW-T) (Experimental): randomized to STRW-T intervention
  Interventions: Behavioral: STRW-T
- Program for the Education and Enrichment of Relational Skills - Telehealth (PEERS-T) (Active Comparator): randomized to PEERS-T intervention
  Interventions: Behavioral: PEERS-T

INTERVENTIONS:
Behavioral: STRW-T — The STRW-T intervention consists of 15 weekly caregiver group sessions and caregiver-teen dyad sessions delivered via Zoom. The targeted daily living skills (DLS) have been identified and refined through our prior studies and include: Morning routine, laundry, kitchen/cooking, grocery shopping, and money management. Evidence-based strategies are utilized to facilitate acquisition, mastery, and generalization of specific DLS at home and in the community. During dyad sessions, teens will work on DLS in their home environment and will receive coaching and instruction from both their caregiver and the therapist. During caregiver group sessions, the therapist will discuss the content of dyad sessions and engage in problem solving with each caregiver (e.g., using and fading rewards, implementing strategies to increase success, teen motivation/buy-in).
  Arms: Surviving and Thriving in the Real World - Telehealth (STRW-T)
Behavioral: PEERS-T — PEERS-T is a 15-week intervention with concurrent caregiver and teen group telehealth sessions that target social skills (e.g., building friendships, conversing, dealing with bullying). PEERS-T was chosen as the control because it is one of the few evidence-based interventions for autistic adolescents and does not address daily living skills. PEERS-T is also matched to STRW-T on duration and is clinically meaningful to families.
  Arms: Program for the Education and Enrichment of Relational Skills - Telehealth (PEERS-T)

SUMMARY:
The current study seeks to compare outcomes of a telehealth intervention targeting daily living skills (Surviving and Thriving in the Real World - Telehealth, or STRW-T) intervention to a control group telehealth intervention targeting social skills (Program for the Education and Enrichment of Relational Skills- Telehealth, or PEERS-T). The key endpoint will be change in daily living skills on primary and secondary outcome measures at the end of treatment.

DETAILED DESCRIPTION:
Individuals with high functioning autism spectrum disorder (ASD) are not developing the skills necessary to successfully transition from adolescence to college, employment, and independent living.

Daily living skills (DLS) have been linked to positive adult outcome in individuals with ASD.

Despite the importance of daily living skills to adult outcome, adolescents with high functioning ASD have impaired daily living skills.

A complex set of environmental, individual, and family factors likely affect the ability of adolescents with high functioning ASD to acquire critical daily living skills.

There are currently no evidence-based daily living skills intervention packages for adolescents with high functioning ASD that would prepare them for independence in adulthood.

A total of 192 autistic adolescents between the ages of 15-21 who are in their last 2 years of high school will be randomized to the STRW-T group (n=96) or the PEERS-T control group (n=96). Outcome measures will be assessed at baseline, post-treatment, 6-month follow-up, and 6-month post-high school graduation assessments. Adolescents will meet the following inclusion criteria: (1) a diagnosis of ASD; (2) enrolled in 11th or 12th grade; (3) Intelligence Quotient of greater than or equal to 70; and (4) a DLS deficit on the Vineland-3 interview as reported by caregivers.

Aim 1: Examine the efficacy of STRW-T on DLS compared to a control group (PEERS-T). Hypothesis 1: STRW-T youth will have greater gains on the primary DLS assessment (VABS-3) compared to PEERS-T youth at post-treatment; Hypothesis 2: STRW-T youth will have greater gains on secondary DLS assessments (Adaptive Behavior Assessment System, 3rd Edition, DLS-Goal Attainment Scale, daily phone diaries) compared to PEERS-T at post-treatment.

Aim 2: Evaluate whether the improvement on DLS outcomes by STRW-T are sustained beyond the intervention period. Hypothesis 3: The impact of STRW-T on DLS gains (as assessed by primary and secondary DLS assessments) will be sustained at 6-months post-treatment.

Aim 3: Examine the effects of the STRW-T intervention on outcomes in college, employment, and Quality of Life after high school graduation. Hypothesis 4: STRW-T youth will have better college, employment, and Quality of Life outcomes compared to PEERS-T youth at 6-months post-high school graduation.

ELIGIBILITY:
Inclusion Criteria:

* in the last 2 years of high school, or deferring graduation
* diagnosis of ASD based on clinical judgement and/or meeting the cut-off score on the Autism Diagnostic Observation Schedule, 2nd Edition
* full scale IQ of 70 or above as measured by the Wechsler Abbreviated Scale of Intelligence, 2nd Edition
* deficient Daily Living Skills as assessed by the Vineland Adaptive Behavior Scales, 3rd Edition - at least 1 of the 3 Daily Living Skills subdomains is at least 15 points below their full scale IQ

Exclusion Criteria:

* significant aggressive behaviors or mental health issues that require treatment out of the scope of the current intervention.
* if the adolescent has already completed the social skills group (PEERS), either at Cincinnati Children's or in another setting, unless it has been a significant amount of time since they did the PEERS group (2-3 years, or up to the discretion of the PI).

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales, 3rd Edition | 4 months
  The VABS-3 is a well-established standardized measure of adaptive behavior that assesses skills in the Communication, Daily Living Skills, and Socialization domains. The DLS domain is comprised of the Personal, Domestic, and Community subdomains and has items that directly correspond to goals being targeted in the STRW intervention.
  Subdomain v-scale scores: 1 to 24. Domain and Adaptive Behavior Composite Standard Scores: 20 to 140. The higher the score, the better the adaptive level. V-scale scores have a mean of 15 and standard deviation (SD) of 3. Standard scores have a mean of 100 and SD of 15.

SECONDARY OUTCOMES:
Adaptive Behavior Assessment System, Third Edition | 4 months
  The ABAS-3 Adult Other measure is a respondent report measure that assesses adaptive behavior in the conceptual, practical, and social domains. The Practical domain standard score summarizes performance across the Community Use, School Living, Health and Safety, and Self-Care skill areas. The standard score is calculated based on the sum of scaled scores for each of the skill areas. Scaled scores range from 1 to 19, with the average score being between 8-12. The standard scores typically range from 40 to 120, with a mean of 100 and a standard deviation of 15. Higher scores equate to better adaptive skills.

CONTACTS AND LOCATIONS:
Overall Officials: Amie Duncan, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - University of North Carolina - Chapel Hill, Carrboro, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No